CLINICAL TRIAL: NCT03132558
Title: Contrast Induced Acute Kidney in Patients With Acute Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hai-Bin Shi, Professor, Nanjing Medical University
Other Study IDs: AISAKI001
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Contrast Media

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CTA: Patients with AIS only receieved cerebral CTA exam.
  Interventions: Drug: Radiopaque Media
- CTA+DSA: Patients with AIS receieved cerebral CTA, followed by endovascular treatment with the guidence of digital substration angiography (DSA).
  Interventions: Drug: Radiopaque Media

INTERVENTIONS:
Drug: Radiopaque Media

SUMMARY:
Computed tomographic angiography (CTA) is recommended for identifying eligible patient with acute ischemic stroke (AIS) to receieve endovascular treatment. We are going to conduct this prospective corhot study to observe if sequential use contrast in CTA examination and in endovascular treatment will cause acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are suspected with AIS.
* Non-contrast head CT excludes intracranial hemorrhage.

Exclusion Criteria:

* Lacking of pre-CTA Creatinine
* Lacking of post-angiography Creatinine with 24-48 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are suspected with AIS. Non-contrast head CT excludes intracranial hemorrhage. Patients who receieve CTA or CTA+DSA will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Creatinine | within 24h to 48h
  Contrast-induced acute kidney injury was defined as a relative increase of 25% or an absolute increase of 0.3 mg/dL (28.2mol/L) in the serum creatinine level at 48 hours following angiography

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia ZY, Wang SX, Zhao LB, Cao YZ, Shi HB, Liu S. Risk of Acute Kidney Injury with Consecutive, Multidose Use of Iodinated Contrast in Patients with Acute Ischemic Stroke. AJNR Am J Neuroradiol. 2019 Apr;40(4):652-654. doi: 10.3174/ajnr.A5959. Epub 2019 Jan 24. PMID 30679214